CLINICAL TRIAL: NCT00653146
Title: Effects of Mindfulness-Based Stress Reduction (MBSR) on Immune Response to HPV
Brief Title: The Effects of MBSR in Improving Immune Response to Human Papillomavirus in Patients With Cervical Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carolyn Fang, PhD, Principal Investigator, Fox Chase Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000590603; 06851 (Other: Fox Chase Cancer Center); R01CA125069 (NIH)
Record Dates: First submitted 2008-04-03; First posted 2008-04-04 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; psychosocial effects of cancer and its treatment; human papilloma virus infection; atypical squamous cells of undetermined significance; low-grade squamous intraepithelial lesion
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Papillomavirus Infections; Atypical Squamous Cells of the Cervix; Squamous Intraepithelial Lesions | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based stress reduction (Experimental): The MBSR program includes meditation techniques, body scan, awareness of breathing, mindful yoga, eating meditation, and walking meditation, and meets for 2 hours, once weekly for 8 weeks.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Healthy Lifestyles Program (Placebo Comparator): The Healthy Lifestyles Program includes information on nutrition and physical activity, and meets for 2 hours, once weekly for 8 weeks.
  Interventions: Behavioral: Healthy Lifestyles

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — In the intervention program, a variety of mindfulness meditation techniques will be taught, including the body scan, awareness of breathing, mindful yoga, eating meditation and walking meditation.
  Other Names: MBSR
  Arms: Mindfulness-based stress reduction
Behavioral: Healthy Lifestyles — In the control condition, information on healthy lifestyles will be presented in a didactic fashion. Session topics include diet and nutrition, physical activity, and healthy behaviors to prevent cardiovascular disease and cancer.
  Arms: Healthy Lifestyles Program

SUMMARY:
RATIONALE: Mindfulness-based stress reduction (MBSR) may reduce patient stress and improve quality of life. It is not yet known whether mindfulness-based stress reduction is effective in improving immune response to human papillomavirus in patients with cervical dysplasia.

PURPOSE: This randomized clinical trial is studying whether mindfulness-based stress reduction (MBSR) or a general diet and physical activity program has any effects on immune response to human papillomavirus in patients with cervical dysplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the effects of a standardized mindfulness-based stress reduction (MBSR) intervention versus a diet and physical activity program on psychosocial well-being (e.g., perceived stress and quality of life) at post-intervention and subsequent follow-up time points.
* To evaluate the effects of an MBSR intervention versus a diet and physical activity program on specific immune response to HPV (i.e., T-cell proliferative response to HPV16 and intracellular cytokine expression of HPV-stimulated T-cells) at post-intervention and follow-up time points.
* To examine the extent to which changes in psychosocial well-being mediate the effects of the intervention on HPV-specific immune response.
* To explore potential mechanisms of action (e.g., self-regulation, expectancies) that are proposed to be responsible for producing intervention effects on psychosocial well-being.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo a mindfulness-based stress reduction intervention (including meditation techniques, body scan, awareness of breathing, mindful yoga, eating meditation, and walking meditation) for 2 hours, once weekly for 8 weeks.
* Arm II: Patients undergo a diet and physical activity program for 2 hours, once weekly for 8 weeks.

In both arms, questionnaires measuring psychosocial factors, demographics, and behavioral risk factors are administered to patients at baseline, within 2 weeks of completing the 8-week programs, and then at 6 and 12 months. Treatment continues in the absence of developing cervical cancer.

Blood is collected for immunologic assays. HPV status and subtype is evaluated in cervical specimens using standard and real-time PCR techniques. Quality of Life is evaluated at baseline, post-intervention, and at 6 and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Referred for a colposcopy following an abnormal Pap smear test result

  * Atypical squamous cells of undetermined significance/positive for human papilloma virus or mild to moderate dysplasia
  * Referred for a second opinion OR patient of record within the medical practice who is undergoing routine recommended follow-up
* Recruited from Fox Chase Cancer Center or Thomas Jefferson University Hospital
* No history of cervical cancer
* No evidence of present invasive carcinoma

PATIENT CHARACTERISTICS:

* Must be able to read and/or communicate in English
* Not pregnant
* No known HIV positivity
* No psychiatric disorder or other disorder that would preclude informed consent

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2007-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Comparison of indices of psychosocial well-being between the mindfulness-based stress reduction (MBSR) and control groups | baseline, post-intervention, 6 months, and 12 months

SECONDARY OUTCOMES:
Comparison of the MBSR and control groups on measures of HPV-specific immune response | baseline, post-intervention, 6 months, and 12 months
Correlation of variations in psychosocial factors (e.g., perceived stress, cancer-related distress, QOL) between treatment group (MBSR vs. attention control) and immunologic outcomes | baseline, post-intervention, 6 months, and 12 months
Effect of treatment group and process variables on psychosocial well-being | baseline, post-intervention, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Fang, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania